CLINICAL TRIAL: NCT07212647
Title: Home-Based Strategies for Knee Osteoarthritis: Comparative Effectiveness of Exercise and Topical Therapy in a Randomized Controlled Trial
Brief Title: Home-Based Strategies for Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sezen Karaborklu Argut, Dr., assistant professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 132409382161
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Knee Osteoarthritis; Knee Osteoarthritis (Knee OA)
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Psychotherapy, Group

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Exercise Group (Experimental): Each subject in the home exercise group will receive a video-based protocol of exercises for knee osteoarthritis to perform at home.
  Interventions: Other: Home Exercise Group
- Topical Therapy Group (Active Comparator): Each subject in the topical therapy group will apply topical gel to anterior, medial, and lateral aspects of the knee at home.
  Interventions: Other: Topical Therapy Group

INTERVENTIONS:
Other: Home Exercise Group — Patient education + structured, video-based home exercise program Participants instructed to perform exercises 5 days per week for 6 weeks Adherence monitored via logs and telephone follow-up at week 3
  Arms: Home Exercise Group
Other: Topical Therapy Group — Patient education + 1.5% diclofenac sodium gel Participants applied gel to anterior, medial, and lateral aspects of the knee, once daily, without massage techniques, for 6 weeks
  Arms: Topical Therapy Group

SUMMARY:
Knee osteoarthritis (KOA) is a common chronic joint condition leading to pain, functional limitations, and reduced quality of life. This randomized controlled trial aims to evaluate and compare the effectiveness of a structured home-based exercise program versus topical diclofenac sodium therapy in improving pain, functional outcomes, and health-related quality of life among adults with early-stage KOA. The results are intended to provide evidence on the optimal components of home-based conservative management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-70 years
* Diagnosed with Kellgren-Lawrence grade I-II knee osteoarthritis
* Ability to provide written informed consent

Exclusion Criteria:

* Advanced KOA (Kellgren-Lawrence grade IV) requiring arthroplasty
* Prior knee surgery within the past year
* Intra-articular injections within the last 3 months
* Neurological, rheumatological, or systemic conditions affecting mobility
* Inability to comply with study procedures

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline
  Pain intensity will be measured using an 11-point numeric pain rating scale, with 0 indicating no pain and 10 indicating the worst pain conceivable. Patients will be asked to rate their knee pain's severity with a number between 0 and 10 using this scale. The minimum clinically important difference (MCID) of this validated pain scale is accepted as >2.
Numeric Pain Rating Scale (NPRS) | Six-week
  Pain intensity will be measured using an 11-point numeric pain rating scale, with 0 indicating no pain and 10 indicating the worst pain conceivable. Patients will be asked to rate their knee pain's severity with a number between 0 and 10 using this scale. The minimum clinically important difference (MCID) of this validated pain scale is accepted as >2.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline
  The assessment of functional difficulty will be measured the WOMAC index. The total score of the WOMAC ranges from 0 to 100 (lower scores representing lower level of disability), and the MCID was reported as 12 points.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Six-week
  The assessment of functional difficulty will be measured the WOMAC index. The total score of the WOMAC ranges from 0 to 100 (lower scores representing lower level of disability), and the MCID was reported as 12 points.
12-Item Short Form Survey (SF-12) | Baseline
  The assessment of health-related quality of life will be measured the 12-Item Short Form Survey (SF-12). The SF-12 physical and mental scores (range 0 to 100, representing worst to best; MCID of 5) was used to evaluate health-related quality of life
12-Item Short Form Survey (SF-12) | Six- week
  The assessment of health-related quality of life will be measured the 12-Item Short Form Survey (SF-12). The SF-12 physical and mental scores (range 0 to 100, representing worst to best; MCID of 5) was used to evaluate health-related quality of life

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpaşa Faculty of Health Science, Istanbul, Buyukcekmece
  - Sezen Karaborklu Argut, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided